CLINICAL TRIAL: NCT03539783
Title: Identification of Pediatric Acute Respiratory Distress Syndrome Subtypes by Bronchial and Nasal Epithelial Transcriptomics
Brief Title: Identifying PARDS Endotypes
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Society of Critical Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_PARDSEndo_001
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Distress Syndrome; Respiratory Distress Syndrome, Adult
Keywords: Endotype; Pediatric Acute Respiratory Distress Syndrome; Gene Expression; Transcriptomics
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA and DNA from brushing specimens. Serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PARDS: Children <18 years of age with PARDS and expected duration of hospitalization seven days or greater.
  Interventions: Diagnostic Test: Respiratory epithelial cell brushing
- Control: Children <18 years of age without PARDS or other lung disease and expected duration of hospitalization 7 days or greater.
  Interventions: Diagnostic Test: Respiratory epithelial cell brushing

INTERVENTIONS:
Diagnostic Test: Respiratory epithelial cell brushing — At specified time points, nasal brushings will be performed to obtain RNA.

SUMMARY:
Pediatric acute respiratory distress syndrome (PARDS) is a severe and diffuse lung injury that is a common cause of admission and mortality in the pediatric intensive care unit (PICU). PARDS can be secondary to many different causes, and there are few therapies that have been shown beneficial in PARDS. This study seeks to identify important PARDS subtypes using gene expression profiling of bronchial epithelial cells from control and PARDS subjects.

DETAILED DESCRIPTION:
Enrolled subjects will have nasal brushings collected at days 1, 3, 7, and 14 of intubation with collection of serum at these same time points. Brushing RNA will be processed by mRNA-Seq for gene expression analysis and compared to previously published serum biomarkers (interleukin-8, advanced glycosylation end-product specific receptor, and angiopoietin-2) to assess correlation and ability to discriminate PARDS endotypes. Changes in gene expression over time will be assessed to define a PARDS recovery gene expression signature, and correlation between bronchial and nasal gene expression will be determined.

ELIGIBILITY:
Inclusion Criteria:

All potential participants must:

1. Be aged zero to 18 years (both control and ARDS, not age matched)
2. Be admitted to the PICU with expected duration of hospitalization 7 days or greater.

ARDS patients must:

1. Have acute changes in chest x-ray (CXR)
2. Have a known or suspected insult within the prior 7 days that is consistent with ARDS
3. Have an oxygenation index (OI) of 4 or greater or and oxygen-sat index (OSI) of 5 or greater

   1. OI = mean airway pressure X fraction inspired oxygen (FiO2) / arterial oxygen partial pressure (PaO2)
   2. OSI = mean airway pressure X FiO2 / oxyhemoglobin saturation (SpO2) with sat <= 97%.

Exclusion Criteria:

1. Have a baseline oxygen requirement of 2 liters of oxygen or greater at home
2. Have disruption of the nasal passages
3. Have a history of excessive bleeding or known bleeding disorders
4. Be at high risk of bleeding
5. Have a do not resuscitate (DNR) or Limited Resuscitation Order

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Control subjects will be patients admitted to the PICU for non-lung injury related conditions.
  PARDS subjects will be intubated patients with PARDS in the PICU.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Identification of PARDS Endotypes | 6 years
  Use of unbiased cluster analysis of gene expression to identify subtypes in PARDS

SECONDARY OUTCOMES:
Lung Recovery Gene Expression Profile | 6 years
  Determination of pathways and processes that differentiate PARDS recovery from non-recovery as assessed by improvement in oxygenation.
Correlation of Nasal and Bronchial Gene Expression | 6 years
  Similarity analysis of bronchial and nasal gene expression in subjects undergoing bronchoscopy to determine whether nasal can be used as a surrogate for bronchial
Correlation of Endotypes with Lung Cell-specific Biomarkers | 6 years
  Matching PARDS endotypes with published markers of hyperinflammatory, microvascular-injury predominant, and distal lung epithelial cell-predominant injury

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Standage, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Study info will be shared with interested investigators on a case by case basis. Microarray data will be posted on an archive such as GeoDatasets but we are unclear how correlative clinical and serum biomarker data would be shared.

REFERENCES:
- [Result] Williams JG, Jones RL, Yunger TL, Lahni PM, Yehya N, Varisco BM. Comparison of 16 Pediatric Acute Respiratory Distress Syndrome-Associated Plasma Biomarkers With Changing Lung Injury Severity. Pediatr Crit Care Med. 2024 Jan 1;25(1):e31-e40. doi: 10.1097/PCC.0000000000003311. Epub 2023 Jun 29. PMID 37382480
- [Result] Williams JG, Joshi R, Haslam D, Yehya N, Jones RL, Paranjpe A, Pujato M, Roskin KM, Lahni PM, Wong HR, Varisco BM. Multi-omic characterization of pediatric ARDS via nasal brushings. Respir Res. 2022 Jul 9;23(1):181. doi: 10.1186/s12931-022-02098-3. PMID 35804409